CLINICAL TRIAL: NCT01932905
Title: Deep rTMS in Central Neuropathic Pain Syndromes
Acronym: DRTMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Daniel Ciampi Araujo de Andrade, MD, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RGDCA-02
Record Dates: First submitted 2013-08-27; First posted 2013-08-30 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Pain; Spinal Cord Injury; Post Stroke Pain
Keywords: deep repetitive transcranial magnetic stimulation; chronic pain; assessment; neuropathic pain; central pain; treatment
MeSH Terms: conditions — Pain; Spinal Cord Injuries; Chronic Pain; Neuralgia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- deep rTMS-active doble coil (Active Comparator): patients undergoing of deep rTMS real with doble coil
  Interventions: Device: deep rTMS
- deep rTMS-sham (Sham Comparator): patients undergoing to placebo deep rTMS
  Interventions: Device: deep rTMS
- deep rTMS-active: H-coil (Active Comparator): patients undergoing of deep rTMS real with H-coil
  Interventions: Device: deep rTMS

INTERVENTIONS:
Device: deep rTMS — Patients undergoing of repetitive transcranial magnetic stimulation for treatment of central pain

SUMMARY:
Pain affects up to 30% of the general population. In particular, neuropathic pain (NeP) is caused by lesion or desease affecting peripheral or central somatosensory pathways and affects 7% of the adult population. Despite the availability of evidence based pharmacological and surgical treatment for NeP, about 50% of patients remais symptomatic despite best medical treatment. Some neuropathic pain syndromes are specially refractory. In particular, central NeP is caused by disease or lesion to central structures involves in somatosensory integration of nociceptive information is non-responsive to drugs usually employed in other NeP syndromes. Classical neuromodulatory techniques such as conventional repetitive Transcranial Magnetic Stimulation aiming at the motor of prefrontal cortices are ineffective to relieve pain in this population. Recently new technology advances have made possible non-invasive stimulation of deeper cortical targets. Some of them are activelly involved in the integration of the perception of pain, such as the anterior cingulate cortex or the posterior insula. The aim this study is to treat 90 patients with central pain (post stroke pain, spinal cord lesions after trauma or demyelinizating diseases) under best medical pharmacological treatment in three different conditions: AAC (n= 30 with the H-Coil), Superior Posterior Insula (SPI) n=30 cooled double cone coil double cool coil, and sham(n=30). Each patients will undergo daily stimulation for a week, then weekly stimulations for 3 months (total of 17 sessions). The main study outcome is pain relief at the last stimulation week (visual-analogic scale). Secondary end-points are changes in the McGill Pain Questionnaire, Neuropathic Pain Symptom Inventory, DN4 questionnaire, SF -36, brief pain inventory and cognitive assessment including the trail making test A and B, Strrop color interference test, and subscalles from the CERAD. All patients will undergo quantitative sensory test and measurements of cortical excitability over M1 before and after to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed term of informed consent
* central pain

Exclusion Criteria:

* Trauma of Skull, epilepsy don't treated,
* Use of medications decrease the seizure threshold
* Patients in use of drugs, how cocaine and alcohol
* neurosurgical clips, pacemakers, increased intracranial pressure (risk of sequelae after seizure)
* Pregnant or lacting women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in baseline of Pain | base line (moment of inclusion) and end of each session rTMS (4X in three months)
  assessing by verbal analog scale (VAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo (HC/FMUSP), São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Galhardoni R, Aparecida da Silva V, Garcia-Larrea L, Dale C, Baptista AF, Barbosa LM, Menezes LMB, de Siqueira SRDT, Valerio F, Rosi J Jr, de Lima Rodrigues AL, Reis Mendes Fernandes DT, Lorencini Selingardi PM, Marcolin MA, Duran FLS, Ono CR, Lucato LT, Fernandes AMBL, da Silva FEF, Yeng LT, Brunoni AR, Buchpiguel CA, Teixeira MJ, Ciampi de Andrade D. Insular and anterior cingulate cortex deep stimulation for central neuropathic pain: Disassembling the percept of pain. Neurology. 2019 Apr 30;92(18):e2165-e2175. doi: 10.1212/WNL.0000000000007396. Epub 2019 Apr 5. PMID 30952795